CLINICAL TRIAL: NCT06565962
Title: 'The Effect of Virtual Reality Use on Disaster Literacy, Disaster Readiness and Disaster Resilience in Adults Living in Rural Areas: A Randomised Controlled Study
Brief Title: The Effect of Virtual Reality Use on Disaster Literacy, Disaster Readiness and Disaster Resilience
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: FATOŞ UNCU (Other)
Responsible Party: Sponsor-Investigator, FATOŞ UNCU, assistant professor, Firat University
Organization: Firat University (Other)
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Prevention
Other Study IDs: FU-SBF-FU-03
Record Dates: First submitted 2024-08-20; First posted 2024-08-22 (Actual); Last update posted 2025-08-12 (Actual); Status verified 2025-08

CONDITIONS: Public Health Nursing
Keywords: Virtual Reality; Disaster Literacy; Disaster Resilience
MeSH Terms: interventions — Control Groups

STUDY DESIGN:
Intervention Model Description: parallel group 1:1 single blind randomised controlled experimental study
Who Masked: Participant
Masking Description: The research will be conducted in a randomised controlled experimental design. The participants randomly assigned to the groups will first be administered data collection forms as a pre-test. Then, the experimental group will be made to watch the training videos prepared by AFAD on disaster preparedness, disaster moment and post-disaster by using virtual reality goggles. Then, data collection for the post-test will be carried out from both groups. After a 3-month follow-up period, follow-up test questionnaires will be collected from both groups. No intervention will be made to the control group. Personal information form, disaster literacy scale, disaster preparedness scale and disaster resistance scale will be used to collect the research data.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Education group (Experimental): Participants randomly assigned to groups will first be given data collection forms as a pre-test. Then, the experimental group will be given an 8-week disaster risk reduction programme. They will watch PowerPoint presentations prepared by researchers and training videos prepared by AFAD on disaster preparedness, disaster response and post-disaster issues using virtual reality glasses. Subsequently, data collection for the post-test will be conducted for both groups. After a three-month follow-up period, follow-up test surveys will be collected from both groups.
  Interventions: Other: Educaiton group
- Control group (Other): The control group will receive standard care. The standard care programme will include brochures and guidance. Personal information form, disaster literacy scale, disaster preparedness scale and disaster resistance scale will be used to collect the research data.
  Interventions: Other: control group

INTERVENTIONS:
Other: Educaiton group — The experimental group will be made to watch training videos prepared by AFAD on disaster preparedness, disaster moment and post-disaster by using virtual reality goggles.
  Arms: Education group
Other: control group — The control group will receive standard care. The standard care programme will include brochures and guidance.
  Arms: Control group

SUMMARY:
Pre-disaster mitigation and preparedness activities are essential to reduce vulnerability in a community and protect people when disasters occur. Although disaster preparedness and protective behaviours have attracted the attention of scholars worldwide, there is no significant study on the preparedness, disaster literacy and disaster resilience of rural households. The aim of this study is to examine the effect of virtual reality use on disaster literacy, disaster preparedness and individual disaster resilience in adults living in rural areas.

DETAILED DESCRIPTION:
In recent years, there has been a significant increase in the number of natural disasters and the loss of life and property caused by disasters in the world and in Turkey. Turkey is a country where tectonic strata are commonly found. Besides, it has various natural disaster risks considering its geological features, topography and meteorological conditions. According to the statistics of the Disaster and Emergency Management Presidency (AFAD) for 2022, the natural disaster events that occurred in 2022 were as follows: 18 avalanches, 21,054 earthquakes, 859 landslides, 137 rock falls, 13 sinkholes, 450 floods/floods and 451 others, totalling 22,982. Considering the high physical and social vulnerability of Turkey, these disasters cause a high number of deaths, injuries and material losses. The solution to minimise the negative impacts of disasters is to be prepared for future disasters. For this reason, there is a need for raising awareness of the society about disasters and disaster risk avoidance skills known as disaster literacy. Disaster literacy is defined as the degree to which individuals read, understand and use information to make informed decisions and follow instructions in the context of mitigation, preparation, response and recovery. In the last decade, virtual reality-based training in disaster preparedness has been increasingly recognised as an important and new alternative to the traditional methods of real-life drills and tabletop exercises. Many studies have described various applications of virtual reality in disaster training. In 2001, Freeman et al. published the use of a virtual reality patient simulation system to teach emergency response skills to US Navy medical personnel. In 2007, a virtual simulation-enhanced triage training for Iraqi medical personnel was described. The following year, immersive simulation for training first responders to mass casualty incidents,mass casualty triage skills using immersive three-dimensional virtual reality, and critical care skills during mass casualty drills. The equivalence of VR simulators with live actor-patient use in directing actions has been demonstrated and simulation for team training and assessment using virtual worlds. In 2009, game-based mass casualty burn training was proposed.In 2011, Cone et al. published a comparison of SALT and SMART triage systems using a virtual reality simulator with paramedic students. Finally, virtual simulation as a teaching method for nursing students has been shown to reinforce learning and improve retention of learning over time.

Pre-disaster mitigation and preparedness activities are essential to reduce vulnerability in a community and protect people when disasters occur. Although disaster preparedness and protective behaviours have attracted the attention of scholars worldwide, there is no significant study on the preparedness, disaster literacy and disaster resilience of rural households. The aim of this study is to examine the effect of virtual reality use on disaster literacy, disaster preparedness and individual disaster resilience in adults living in rural areas.

ELIGIBILITY:
Inclusion Criteria:

* Over 18 years of age
* Not having received structured disaster training before
* Not having any mental problems that prevent them from completing the questionnaires

Exclusion Criteria:

* Participants wants to leave the study
* Incomplete filling of survey forms

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 64 (Actual)
Dates: Start 2024-09-15 (Actual); Primary Completion 2025-01-15 (Actual); Study Completion 2025-02-15 (Actual)

PRIMARY OUTCOMES:
Disaster literacy scale | 3 month
  It is a self-report scale developed by Çalışkan and Üner (2023) to evaluate AFOY in people aged 18-60 years. The scale consists of 61 items and four sub-dimensions: harm reduction, preparation, intervention and improvement. Likert-type scale is graded from 1=very difficult to 5=very easy. There are no reverse items in the scale. The total score that can be obtained from the scale is between 61-305. The high score obtained from the scale shows that the disaster literacy level of individuals is high. In the scale, 0 indicates the lowest AFOY and 50 indicates the highest AFOY. The scale is divided into criteria as 0-<30 points inadequate AFOY, 30-<36 points limited AFOY, 36-<42 points adequate AFOY and 42-50 points excellent AFOY: Scores= (0-<30): inadequate AFOY; (30-<36): limited AFOY; (36-<42): adequate AFOY; (42-50): excellent AFOY. Cronbach's alpha coefficient for internal consistency of the whole scale is α=0.954.

SECONDARY OUTCOMES:
Disaster preparedness scale | baseline (pre test), post test (8 week) and after 3 month
  It was developed by Şentuna and Çakı to determine the preparedness of individuals for disasters. The scale consists of a measurement tool consisting of 13 items and 4 dimensions. The scale consists of four (4) sub-dimensions as 'disaster physical protection', 'disaster planning', 'disaster assistance' and 'disaster warning systems'. There are five items in the 'disaster physical protection' sub-dimension, three items in the 'disaster planning' sub-dimension, three items in the 'disaster relief' sub-dimension and two items in the 'disaster warning systems' sub-dimension. The items in the scale are in 4-point Likert format as '1-Strongly No', '2-No', '3-Yes', '4-Strongly Yes'. The minimum score that can be obtained from the scale is 13 and the maximum score is 52. As the score obtained from the scale increases, the level of disaster preparedness increases. Cronbach Alpha coefficient calculated for the whole scale is 0,82.
Individual Disaster Resilience Scale | baseline (pre test), post test (8 week) and after 3 month
  The scale developed by Şen (2022) consists of 20 items and four sub-dimensions. These sub-dimensions are coping with experience, coping with knowledge, coping with common coping and emotional coping. The scale is Likert 5 type and the questions are scored between 1: strongly disagree and 5: strongly agree. Three items in the scale are reverse coded. The higher the score, the higher the disaster resilience is considered to be

CONTACTS AND LOCATIONS:
Locations (1):
- Firat University, Elâzığ, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No